CLINICAL TRIAL: NCT00459680
Title: Acupuncture and Laser Acupoint Treatment on Hypertension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: John Zhang, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCC-05-06
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension
Keywords: hypertension; acupuncture; laser
MeSH Terms: conditions — Hypertension | interventions — Lasers; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Laser Acupoint (Experimental)
  Interventions: Device: Laser acupoint treatment

INTERVENTIONS:
Device: Laser acupoint treatment — Laser
  Other Names: Laser
  Arms: Laser Acupoint
Procedure: Acupuncture — Needle acupuncture on ST36 and LI11.
  Arms: Acupuncture

SUMMARY:
To determine the effect of acupuncture and laser acupuncture point treatment on hypertensive subjects.

DETAILED DESCRIPTION:
The specific aims of the study are to test the effectiveness of acupuncture and laser acupoint on hypertension. The hypothesis is: the stimulation of a pattern of acupoints with acupuncture and laser will result in significant reductions in blood pressure. The points that are going to be used for the study are: Zusanli (St36), Tianshu (St25), Quchi (LI11).

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 and under 70 years of age with hypertension (blood pressure over 140/90 mmhg).

Exclusion Criteria:

* Individuals with heart, kidney, thyroid disorders, diabetes, chronic disease or illness, neurological diseases, skin or bleeding disorders, and currently taking drugs or medications will not be recruited in the study. A health history questionnaire will be used to screen the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-01 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Pretreatment then at 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD. PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States